CLINICAL TRIAL: NCT06513390
Title: The Development of an Exoskeleton System for Assisting and Enhancing Patients' Mobility.
Brief Title: Development of an Exoskeleton for Patients' Mobility.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vidyasirimedhi Institute of Science & Technology (VISTEC) (Other)
Responsible Party: Principal Investigator, Krongkaew Klaewkasikum, Faculty of Medicine, Ramathibodi Hospital, Mahidol University., Vidyasirimedhi Institute of Science & Technology (VISTEC)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Grant No. I20POM-INT010
Record Dates: First submitted 2024-07-09; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Healthy
Keywords: Exoskeleton; Gait; Kinematics; Temporal spatial; Muscle activity; Oxygen consumption

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- healthys received intelligent mode first (Active Comparator): healthy subjects received exoskeleton with intelligent mode first
  Interventions: Device: Exoskeleton of default mode; Device: Exoskeleton of Intelligent mode
- healthys received default mode first (Placebo Comparator): healthy subjects received exoskeleton with intelligent mode first
  Interventions: Device: Exoskeleton of default mode; Device: Exoskeleton of Intelligent mode

INTERVENTIONS:
Device: Exoskeleton of default mode — Default mode: A standard control system offering a conventional assistive function of Exo-H3.
Device: Exoskeleton of Intelligent mode — Intelligent mode: The adaptive CPG-based control system developed by our researchers from Exo-H3.

SUMMARY:
The goal of this clinical trial is to investigate the performance of a state-of-the-art adaptive CPG-based exoskeleton control system (intelligent mode) under a multi-metric analysis (involving three-dimensional gait analysis, muscle activity, oxygen consumption, user comfort, and exoskeleton performance scores) and comparing it to a standard commercial exoskeleton control system (default mode)

The main question it aims to answer is: Could the adaptive version improve natural walking and essential lower limb motions?

Participants will:

All participants were assigned into two groups to receive an alternate sequence of walking with the intelligent mode or the default mode of the lower-limb exoskeleton Exo-H3 at high and normal speed.

ELIGIBILITY:
Inclusion Criteria:

* healthy Thai adults
* age between 18 and 60 years old
* body mass index between 18.5 and 24.9 kg/m2
* walk independently
* willing to participate in the study

Exclusion Criteria:

* a history of surgery in the back, hip, knee, or ankle area
* previous injury or pain in the hip, knee, or ankle area that would affect walking patterns within the past 6 months
* a history of musculoskeletal or neuromuscular disease such as multiple sclerosis, myasthenia gravis
* a balance disorder
* unable to continue or withdrawal from the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 8 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
gait kinematic of pelvic hip, knee and ankle joint. | 1 day
  The average of pelvic-hip-knee-ankle angles (degrees) in frontal, sagittal and transverse plance were collected by using three dimensions with an eight-camera Motion analysis (Motion Analysis Corporation, Santa Rosa, CA, USA).

SECONDARY OUTCOMES:
Temporal spatial data of velocity | 1 day
  Mean velocity (m/s) was collected by an eight-camera Motion analysis (Motion Analysis Corporation, Santa Rosa, CA, USA).
Temporal spatial data of cadence | 1 day
  Mean cadence (step/min) was collected by an eight-camera Motion analysis (Motion Analysis Corporation, Santa Rosa, CA, USA).
Temporal spatial data of step length, step width, and stride length | 1 day
  Mean of step length(cm), step width(cm), and stride length(cm) were collected by an eight-camera Motion analysis (Motion Analysis Corporation, Santa Rosa, CA, USA).
Temporal spatial data of stance phase and swing phase time | 1 day
  Mean percentage of stance phase and swing phase time were collected by an eight-camera Motion analysis (Motion Analysis Corporation, Santa Rosa, CA, USA).
Muscle activity | 1 day
  Bilateral muscles activities of gluteus medius, gluteus maximus, tensor fascia latae, rectus femoris, bicep femoris, medial gastrocnemius, and tibialis anterior muscles during walking were quantified as root mean square (RMS) in the voltage
Oxygen consumption | 1 day
  VO2 MAX (ml/kg/min) was estimated for the walking trial.
user comfort scores | 1 day
  The wearer's opinion to the device, their perceived change, emotion on self-image, anxiety on security, harm or painful, attachment, and movement were evaluated as the comfort score. Each item rated from a 1 (the least problem) to 5 (the most problem). Sum of total score was 30, and categorized as very comfortable (1-6 points), comfortable (7-17 points), moderately comfortable (18 points), uncomfortable (19-29 points), and uncomfortable at all (30 points). The outcome was measured after completing the walk in each exoskeleton mode.
exoskeleton performance scores | 1 day
  The exoskeletal performance questionnaire comprised 2 domains; pain (walking, climbing stairs, rising from sitting, standing) and difficulty (descending stairs, ascending stairs, rising from sitting, standing, bending to floor, walking on even floor, walking for distance). Each item rated from 1 (minimal issues) to 5 (significant problems). The total performance score was designated as the best performance (1-11 points), good performance (12-13 points), moderate performance (33 point), poor performance (34-54 points), and the worst performance (55 points).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Ramathibodi Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No